CLINICAL TRIAL: NCT06363058
Title: Effect of Combined ES Cycling Training on Individuals With SCA
Brief Title: Electrical Stimulation Cycling Training Effects on SCA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung University (Other)
Responsible Party: Principal Investigator, Ya-Ju Chang, Professor, Chang Gung University
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 201902166B0
Record Dates: First submitted 2024-03-28; First posted 2024-04-12 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Spinocerebellar Ataxia (SCA)
Keywords: Motor Control; Motor Learning; Priming; Excitability
MeSH Terms: conditions — Spinocerebellar Ataxias

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Stage 1: Healthy people (No Intervention): To establish a baseline and ensure reliability, and to develop a training protocol for stage 3.
- Stage 2: Short-term training SCA people (Experimental): Short-term ES Cycling Training
  Interventions: Other: ES Cycling Training
- Stage 2: SCA Control group (No Intervention): Control Group
- Stage 3:Long-term training SCA people (Experimental): Long-term ES Cycling Training
  Interventions: Other: ES Cycling Training
- Stage 3: SCA Control group (No Intervention): Control group

INTERVENTIONS:
Other: ES Cycling Training — Implementing Electrical Stimulation (ES) Cycling combined with priming strategies to enhance motor learning tasks
  Arms: Stage 2: Short-term training SCA people; Stage 3:Long-term training SCA people

SUMMARY:
To focuses on the challenges faced by individuals with spinocerebellar ataxia (SCA), highlighting the major clinical sign of ataxia that affects their stability and ability to perform daily activities, thereby impacting their quality of life. It outlines the concept of neural plasticity, which is the brain's ability to adapt through changes in excitability, and notes that these changes are more enduring in the central nervous system (CNS) than in the peripheral nervous system (PNS). This adaptability, crucial for memory and motor learning, is compromised in SCA patients due to impaired brain areas and pathways. The summary further delves into motor learning, distinguishing between explicit and implicit learning, and points out that SCA patients exhibit deficiencies in procedural learning and cerebellar function. It also introduces the concept of priming as a preparatory mechanism that can enhance the effectiveness of physical therapy by modifying subsequent responses to stimuli. The document suggests that cycling, as an aerobic exercise, could prime the brain for improved blood flow and oxygenation, thereby supporting synaptic plasticity and the release of beneficial neurotrophic factors. Finally, the project aims to deepen the understanding of motor performance and learning mechanisms in SCA patients and apply these insights to clinical rehabilitation strategies.

DETAILED DESCRIPTION:
Ataxia is the major clinical sign of spinocerebellar ataxia (SCA) patients. Increased postural sway and instability during volitional movements appear and hinder SCA patients from performing normal daily life activities and influence quality of life of victims.

Neural plasticity comes from excitability changes. Changes in excitability produced by repetitive activities at synapses maintain a longer time in the central nervous system (CNS) than the changes in the peripheral nervous system (PNS). The long duration of synaptic excitability changes may be linked to memory and motor learning. Neural plasticity could be investigated by several non-invasive instruments, such as Transcranial Magnetic Stimulation (TMS). The excitability is suppressed in SCA patients due to corrupted brain areas and pathways.

Motor learning is the process of obtaining the capability for movement. Motor learning is not merely focusing on changes in performance during practice but also being evaluated during retention and/or transfer. Motor learning can be divided into explicit and implicit learning. One type of implicit learning is the acquisition of motor skills, often referred to as procedural learning. Serial reaction time task (SRTT) is used to describe implicit sequence motor learning. A series of implicit motor sequence learning tasks is to clarify the role and function of the cerebellum. And this function is deficient in SCA patients.

Priming is an unconscious process associated with learning to alter the later response by the proceeding stimulus. Priming is applied to physical therapy; it could result in behavioral change and strengthen the training effect afterward.

Cycling could be an aerobic exercise priming that may help to raise brain blood flow and oxygenation, facilitate synaptic plasticity, augment the release of neurotrophic factors, to transmit neuroendocrine and myokines.

This project will advance the knowledge of the mechanism of motor performance and motor learning in SCA individuals. The result of this project can be applied to the clinical rehabilitation of people with SCA.

ELIGIBILITY:
Health subjects:

Exclusion Criteria:

* Musculoskeletal injuries on legs.
* Osteoporosis.

SCA subjects:

Inclusion Criteria:

- Clinical diagnosis of SCA.

Exclusion Criteria:

* Musculoskeletal injuries on legs
* Osteoporosis.
* Any peripheral or central nervous system injury or disease patients.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 145 (Estimated)
Dates: Start 2022-04-08 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Overall Response Time | Baseline, 2 weeks and 4 weeks
  The sum of reaction time and movement time, providing a complete measure of the time taken from the stimulus presentation to the completion of the response. Unit: Second(s)
Overall Error Rate | Baseline, 2 weeks and 4 weeks
  The total proportion of incorrect responses across a testing session or series of tasks.
Motor Evoked Potentials (MEPs) | Baseline, 2 weeks and 4 weeks
  MEPs are the electrical responses recorded from muscles following stimulation of the motor cortex. They reflect the efficiency of neural transmission from the cortex to the muscle. Unit: millivolts (mV).
Intracortical Facilitation (ICF) | Baseline, 2 weeks, and 4 weeks.
  ICF is measured by applying a pair of TMS pulses with a short interval (e.g., 8-15 ms) where the first (subthreshold) pulse is followed by a second (suprathreshold) pulse, leading to an increased amplitude of the MEP.
Intracortical Inhibition (ICI) | Baseline, 2 weeks, and 4 weeks.
  ICI is measured similarly to ICF but with a shorter inter-stimulus interval (e.g., 1-5 ms), resulting in a suppressed MEP amplitude. This suppression reflects inhibitory processes within the cortex.
Total Scale for the Assessment and Rating of Ataxia (SARA) Score | Baseline, 2 weeks, and 4 weeks.
  To objectively assess ataxia severity across various domains of motor function including gait, stance, sitting, speech disturbance, finger chase, nose-finger test, fast alternating hand movements, and heel-shin slide. Each item is scored individually with a scale that typically ranges from 0 (no ataxia) to a maximum score that depends on the severity and the aspect of ataxia being assessed. The total score ranges from 0 (no ataxia) to 40 (most severe ataxia).
Total Berg Balance Scale (BBS) Score | Baseline, 2 weeks, and 4 weeks.
  To measure an individual's balance abilities through various tasks that mimic daily activities, assessing the risk of falls and overall balance proficiency. The BBS consists of 14 items that evaluate a range of functions including sitting to standing, standing unsupported, transferring, turning to look behind, picking up an object from the floor, and standing on one leg. Each task is rated on a scale from 0 (unable) to 4 (independent), with the total score ranging from 0 to 56. A higher total score indicates better balance and lower fall risk. Scores below 45 are generally indicative of increased fall risk.
Total Time to Complete the Time Up and Go test (TUG test) | Baseline, 2 weeks, and 4 weeks.
  The time, in seconds, it takes for a participant to complete the TUG test from the initial sitting position to returning to the seated position. An older adult who takes ≥12 seconds to complete the TUG is at risk for falling.
Walking Speed | Baseline, 2 weeks, and 4 weeks.
  The time taken by participants to walk a standardized distance, typically expressed in centimeters per second (cm/s).
Step Length | Baseline, 2 weeks, and 4 weeks.
  The linear distance between the two ankles, typically expressed in centimeter(cm).
Step Time | Baseline, 2 weeks, and 4 weeks.
  The duration taken for one complete step, measuring from foot-off of one foot to the next foot-off of the same foot, usually expressed in seconds.

SECONDARY OUTCOMES:
Double Support Time | Baseline, 2 weeks, and 4 weeks.
  The portion of the gait cycle where both feet are in contact with the ground, indicating the transition phase between steps, expressed as a percentage of the gait cycle or in seconds.
Single Support Time | Baseline, 2 weeks, and 4 weeks.
  The duration within the gait cycle when only one foot is in contact with the ground, typically measured in seconds or as a percentage of the total gait cycle
Swing Time | Baseline, 2 weeks, and 4 weeks.
  The portion of the gait cycle where the foot is not in contact with the ground, moving forward to the next step. It is usually expressed as a percentage of the total gait cycle or in seconds.
Stance Time | Baseline, 2 weeks, and 4 weeks.
  The portion of the gait cycle when the foot is in contact with the ground, supporting body weight. It's typically expressed as a percentage of the total gait cycle or in seconds
Cadence | Baseline, 2 weeks, and 4 weeks.
  The number of steps an individual takes per minute, providing an overview of gait speed and rhythm, , expressed as steps per minute.

CONTACTS AND LOCATIONS:
Locations (1):
- Chang Gung University, Taoyuan District, Taiwan